CLINICAL TRIAL: NCT01749917
Title: Therapeutic Intervention in Motor Disorders in Parkinson.
Brief Title: Exercise Intervention and Dexterity in Parkinson
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Assistant professor, Universidad de Granada
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DF0036UG
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Parkinson
Keywords: Parkinson.; Dexterity.; Balance.; Exercises.
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Active Comparator): 30 people are recruited in order to the inclusion criteria for the study. The study include subjects who can complete the assessment battery of tests at the beginning and end in order to perform the control intervention.
  Interventions: Other: Control intervention
- Exercise program group (Experimental): 30 people are recruited, diagnosed with Parkinson attending to the Parkinson Association of Granada aged between 40 and 65 years. No sex differences. The study include subjects who can complete the assessment battery of tests at the beginning and end.
  Interventions: Other: Exercise program

INTERVENTIONS:
Other: Exercise program — Exercise program An brief exercise session including proprioceptive and dexterity activities
  Other Names: Plaster of resistance activities
  Arms: Exercise program group
Other: Control intervention — Active upper limb range of movement exercises for 15 minutes.
  Arms: Control group

SUMMARY:
The investigators conducted an intervention based in proprioceptive exercises and balance tasks. The investigators also carried out a brief intervention in manual dexterity.

The study hypothesis is that a brief intervention in upper extremities and a exercise program can increase functionality in Parkinson.

DETAILED DESCRIPTION:
Motor symptoms in Parkinson frequently affect upper extremities. This has been associated in previous studies with limitation in the performance of activities of daily living and, consequently, with a decrease in quality of life. The possibility that a brief intervention improves eye-hand dexterity in Parkinson's, may be a therapeutic option to improve the performance of activities of daily living. The investigators also conducted an intervention based in proprioceptive exercises and balance tasks to improve functionality.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with Parkinson attending to the Parkinson Association of Granada.
* Subjects who can complete the assessment battery of tests at the beginning and at the end of the study.

Exclusion Criteria:

* Auditive and visual disturbances.
* Cognitive problems.
* Psychiatric pathology.
* Sensorial disturbances.
* Traumatic pathology of the hand.
* Concomitant neurological conditions.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Manual dexterity | baseline, 6 months
  Change from baseline to postintervention in dexterity. This is assessed using the Purdue Pegboard Test.
  The Purdue pegboard test is a timed physical test used to measure manual dexterity. Test subjects are asked to place small pins into holes in the pegboard using a specific hand and following a specific process.

SECONDARY OUTCOMES:
Grip strength | baseline, 6 months
  Grip strength is measured using a Jamar dynamometer with a standard protocol allowing three attempts on each side. During each measurement, patients were sitting with their shoulder adducted and elbow flexed to 90°. The maximum value achieved from all six attempts was used in analyses.
  Kg/cm2
Pressure pain measure | baseline, 6 months.
  The pressure pain threshold for each site (three points in upper extremities) is assessed using the pressure algometer. All assessments were made by the same investigator. All the subjects were trained to familiarize the subjects with the pressure algometry procedure before the measures in an anatomical site different from the chosen sites for this study.
Nervous assessment | baseline, 6 months.
  Neurodynamic tests are used in upper extremities. It moves most of the nerves between the neck and hand, including the median nerve, radial and ulnar, brachial plexus, spinal nerves and cervical nerve roots.
  The patient is placed supine position. It is measured with a goniometer.
Risk of falls. | baseline, 6 months.
  The risk of falls is measured with the timed up and go. It measures in seconds, the time taken by an individual to stand up from a standard arm chair,walk a distance of 3 meters, turn, walk back to the chair, and sit down.

CONTACTS AND LOCATIONS:
Overall Officials: M. Carmen Valenza, PH MD, Principal Investigator — Department of Physical Therapy. University of Granada.
Locations (1):
- Faculty of Health Sciences. University of Granada., Granada, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mateos-Toset S, Cabrera-Martos I, Torres-Sanchez I, Ortiz-Rubio A, Gonzalez-Jimenez E, Valenza MC. Effects of a Single Hand-Exercise Session on Manual Dexterity and Strength in Persons with Parkinson Disease: A Randomized Controlled Trial. PM R. 2016 Feb;8(2):115-22. doi: 10.1016/j.pmrj.2015.06.004. Epub 2015 Jun 14. PMID 26079867